CLINICAL TRIAL: NCT02954146
Title: Mobile Health Application for Family and Behavioral Health Provider Communication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InferLink Corporation (Industry)
Collaborators: Duke University (Other); University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00069014
Record Dates: First submitted 2016-10-24; First posted 2016-11-03 (Estimated); Last update posted 2018-03-08 (Actual); Status verified 2018-03

CONDITIONS: Posttraumatic Stress Disorder; Anger
Keywords: Veterans; Posttraumatic Stress Disorder; Anger; Behavioral Health; Mobile Health Technology
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBT only (Active Comparator): Veterans will receive 12 weekly individual cognitive behavioral therapy (CBT only) sessions for anger management.
  Interventions: Behavioral: Connectd mobile application
- CBT + Connectd mobile health app (Experimental): Veterans will receive 12 weekly individual cognitive behavioral therapy (CBT) sessions for anger management. In addition, veterans in this group will also receive instructions for using Connectd mobile health app with a family member or friend that will provide data for the CBT clinician.
  Interventions: Behavioral: Connectd mobile application

INTERVENTIONS:
Behavioral: Connectd mobile application — Connectd is a mobile application that collects and automatically analyzes input from patients with PTSD/TBI, as well as their families, for clinician review. The app will aggregate patient and family input on current issues, relationship stressors, and situational stressors to better focus (personalize) treatment as well as to more efficiently and accurately understand key factors and root causes. In addition, the app provides informational resources for veterans and family regarding treatment options and mental health supports.

SUMMARY:
The purpose of this study is to examine feasibility, tolerability, utilization, and effectiveness of using the SupportTeam mobile application in the context of Cognitive Behavioral Therapy (CBT) for veterans with PTSD.

DETAILED DESCRIPTION:
Purpose: we will examine feasibility, tolerability, utilization, and effectiveness of using the SupportTeam mobile application in the context of Cognitive Behavioral Therapy (CBT) for veterans with PTSD.

Participants: (N=100) 50 veterans who have served in the military since October 2001 and have PTSD with anger problems; and 50 collateral family members/close friends above the age of 18.

Procedures (methods): All Veterans with PTSD will receive a 12 session standard CBT for anger. Veterans in the intervention group will additionally receive instructions for using SupportTeam with a family member or friend that will provide data for the CBT clinician. Veterans in the control group will receive the CBT sessions, but will not receive the SupportTeam mobile application.

ELIGIBILITY:
Inclusion Criteria:

For Veteran:

* Age 18 or older
* Served in a branch of the US military since October, 2001
* Meets DSM-5 criteria for current PTSD as measured by the Clinician-Administered PTSD Scale for DSM-5 (CAPS-5);
* Reports at least one episode of anger or irritability in the past week;
* Has and regularly uses an iOS (iPhone 5s or higher with iOS 8 or higher) or Android (with 4G network and Android 4.1 or higher) smartphone with a data plan;
* Has a family member or friend who also has and uses a smartphone with a data plan and agrees to participate in the study.
* Is able and willing to attend 12 weekly sessions at Duke Psychiatry offices within normal business hours (M-F 8:00-5:00)

For Collateral:

* 18 years old or older
* Has and regularly uses an iOS (iPhone 5s or higher with iOS 8 or higher) or Android (with 4G network and Android 4.1 or higher) smartphone with a data plan;
* Has a family member or friend who meets the veteran inclusion criteria and agrees to participate in the study.

Exclusion Criteria, Veteran:

- Is currently participating in, or is scheduled to participate in a manualized psychosocial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-03-05 (Actual); Study Completion 2018-03-05 (Actual)

PRIMARY OUTCOMES:
Working Alliance Inventory (Short Form, Therapist) | 12 weeks
  Documents perspectives of therapist-client relationship
Participant Treatment Participation | 12 weeks
  Number of weekly sessions attended by participants
Working Alliance Inventory (Client) | 12 weeks
  Documents perspectives of therapist-client relationship
PTSD Knowledge Scale | 12 weeks
  Measures general knowledge about PTSD
Zarit Burden Interview | 12 weeks
  Measures stress felt by caregivers

SECONDARY OUTCOMES:
Dimensions of Anger Reactions | 12 weeks
  Measure of anger disposition towards others
Clinician-Administered PTSD Scale for DSM5 (CAPS 5) | Past month
  Assessment of PTSD symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Eric Elbogen, PhD, Principal Investigator — Duke; Greg Barish, PhD, Study Chair — InferLink Corporation; Patricia E Lester, MD, Study Chair — University of California, Los Angeles
Locations (1):
- Duke University, Department of Psychiatry, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No